CLINICAL TRIAL: NCT00437294
Title: A Double-Blind, Randomized, Phase 2 Trial of Capecitabine Plus Enzastaurin Versus Capecitabine Plus Placebo in Patients With Metastatic or Recurrent Breast Cancer Previously Treated With an Anthracycline and a Taxane
Brief Title: Enzastaurin in Combination of Capecitabine to Treat Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10536; H6Q-MC-S035 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — enzastaurin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capecitabine + Enzastaurin (Experimental)
  Interventions: Drug: enzastaurin; Drug: capecitabine
- Capecitabine + Placebo (Placebo Comparator)
  Interventions: Drug: placebo; Drug: capecitabine

INTERVENTIONS:
Drug: enzastaurin — 1125 milligrams (mg) loading dose then 500 mg, oral, daily, 21-day cycles until progressive disease
  Other Names: LY317615
  Arms: Capecitabine + Enzastaurin
Drug: placebo — oral, daily, 21-day cycles until progressive disease
  Arms: Capecitabine + Placebo
Drug: capecitabine — 1250 mg/m^2, BID, days 1-14 of each 21-day cycle until progressive disease

SUMMARY:
The purpose of this study is to determine whether the combination of enzastaurin and capecitabine is more effective than the combination of placebo and capecitabine in treating participants with breast cancer who were previously treated with an anthracycline and a taxane.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with metastatic or recurrent breast cancer.
* Have been previously treated with both an anthracycline and a taxane.
* Have not received more than two prior chemotherapy treatment programs.
* Have stopped any antitumoral hormonal treatment before you enroll in this study.
* Have a negative pregnancy blood test if menstruating or capable of becoming pregnant. You must use an approved birth control method during the study and for 3 months after stopping study treatment.

Exclusion Criteria:

* Cannot follow the study procedures (for example, you cannot swallow tablets).
* Are receiving another treatment for your cancer.
* Have received another experimental drug in the last 4 weeks.
* Have had serious heart disease within last 6 months.
* Are pregnant or breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Resistencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucumain
- Australia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garran, Australian Capital Territory
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caringbah, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankston, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Subiaco, Western Australia
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avignon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Roche-sur-Yon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Brieuc
- Mexico (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Acapulco
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuernavaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban, South Africa

REFERENCES:
- [Derived] Clemons M, Joy AA, Abdulnabi R, Kotliar M, Lynch J, Jordaan JP, Iscoe N, Gelmon K. Phase II, double-blind, randomized trial of capecitabine plus enzastaurin versus capecitabine plus placebo in patients with metastatic or recurrent breast cancer after prior anthracycline and taxane therapy. Breast Cancer Res Treat. 2010 Nov;124(1):177-86. doi: 10.1007/s10549-010-1152-0. Epub 2010 Sep 3. PMID 20814815
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow reports those participants who discontinued from study drug.
Groups:
- Capecitabine + Enzastaurin: Capecitabine: 1250 milligrams per square meter (mg/m^2), twice daily (BID) on Days 1-14 followed by a 1-week rest period (Days 15-21) for each 21-day cycle until progressive disease.
  Enzastaurin: 1125-milligram (mg) loading dose on Day 1 of Cycle 1, then 500 mg daily on subsequent days to complete 21-day cycles until progressive disease.
- Capecitabine + Placebo: Capecitabine: 1250 mg/m^2, BID on Days 1-14 followed by a 1-week rest period (Days 15-21) for each 21-day cycle until progressive disease.
  Placebo: taken as 4 tablets orally, daily, to complete 21-day cycles until progressive disease.
Period: Overall Study
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo
Started | 43 | 43
Received at Least 1 Dose of Study Drug | 42 | 43
Completed | 0 | 0
Not Completed | 43 | 43
Not completed — Adverse Event | 5 | 4
Not completed — Death | 5 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Progressive Disease | 19 | 23
Not completed — Sponsor Decision | 8 | 9
Not completed — Protocol Violation | 0 | 1
Not completed — Entry criteria not met | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Capecitabine + Placebo: Capecitabine: 1250 mg/m^2, BID on Days 1-14 followed by a 1-week rest period (Days 15-21) for each 21-day cycles until progressive disease.
  Placebo: taken as 4 tablets orally, tablets daily, to complete 21-day cycles until progressive disease.
- Total: Total of all reporting groups
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.73 (10.06) | 52.14 (9.78) | 53.91 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 43 | 85
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 36 | 38 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 31 | 62
  Black or African American | 3 | 0 | 3
  Asian | 2 | 7 | 9
  Hispanic | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 3 | 3 | 6
  Mexico | 3 | 4 | 7
  Argentina | 9 | 7 | 16
  Australia | 11 | 11 | 22
  Canada | 16 | 18 | 34
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — The BMI was reported for 41 participants from each treatment arm. BMI is a measure of body fat based on height and weight that applies to adult men and women.
  kilograms per square meter (kg/m^2) | 27.25 (6.48) | 27.04 (4.95) | 27.14 (5.73)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] — The BSA was reported for 41 participants from each treatment arm. Calculated to express in square meter (m^2).
  square meter (m^2) | 1.73 (0.20) | 1.76 (0.20) | 1.75 (0.20)
Disease Stage [Count of Participants; unit: Participants] — Stage (St) I-small tumor without spread to the axillary lymph nodes (ALN). St II-small to large with or without spreading to nearby ALN, St IIA-no tumor in breast but found in 1-3 ALN; tumor in breast <2.0cm plus spread to ALN; tumor is >2 to 5cm and no spread to ALN. St IIB-tumor >2 to 5cm with spread to 1-3 ALN; tumor is >5 cm with no LN spread. St IIIA- tumor any size with spread to 4-9 ALN or internally mammary LN; the tumor is > 5cm; spread to 1 to 3 ALN. St IIIB-spread to chest and/or skin. St IIIC-spread to 10 or more ALN. St IV and IVB- cancer has spread to other organs of the body.
  Participants
    Stage I | 2 | 3 | 5
    Stage II | 5 | 10 | 15
    Stage IIA | 5 | 5 | 10
    Stage IIB | 6 | 7 | 13
    Stage III | 2 | 5 | 7
    Stage IIIA | 10 | 1 | 11
    Stage IIIB | 7 | 3 | 10
    Stage IIIC | 2 | 7 | 9
    Stage IV | 2 | 2 | 4
    Stage IVB | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from randomization to the first observation of disease progression or death due to any cause. For participants not known to have died as of the data cut-off date and who did not have progressive disease, PFS was censored at the date of last visit with adequate assessment. For participants who received subsequent anticancer therapy (after discontinuation from the study treatment) prior to disease progression or death, PFS was censored at the date of last visit with adequate assessment prior to the initiation of post-discontinuation anticancer therapy.
Time Frame: Randomization to measured progressive disease or death up to 14 months
Population: Intent-to-treat (ITT) population: All randomized participants who received at least 1 dose of study drug.
  Participants censored: Capecitabine + Enzastaurin = 13; Capecitabine + Placebo = 14.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Capecitabine + Enzastaurin: Capecitabine: 1250 milligrams per square meter (mg/m^2), twice daily (BID) on Days 1-14 followed by a 1-week rest period (Days 15-21) for each 21-day cycle until progressive disease.
  Enzastaurin: 1125 1125-milligram (mg) loading dose on Day 1 of Cycle 1, then 500 mg daily on subsequent days to complete 21-day cycles until progressive disease.
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo
Number analyzed (Participants) | 42 | 43
months | 2.79 [2.10 to 4.63] | 4.27 [2.89 to 6.18]
Statistical Analysis 1: Comparison: Capecitabine + Enzastaurin vs Capecitabine + Placebo; Test type: Superiority or Other; p = 0.237, Log Rank — The 1-sided significance level was 0.20

2. Secondary Outcome: Expression of Tumor Markers in Tissue Samples (Tumor Markers and Genes Evaluation)
Description: Protein expression was planned to be measured using an Immunohistochemistry (IHC) assay to determine membrane and cytoplasmic phosphorylated glycogen synthase kinase 3 beta (pGSK3B), nuclear phosphorylated adenosine 3'5'-cyclic monophosphate (cAMP) response-element binding protein (pCREB), cytoplasmic pCREB, protein kinase C beta 2 (PKCB2), cytoplasmic phospho S6 (pS6), and cytoplasmic phosphatase and tensin homolog (PTEN) IHC H-scores. Tumor tissue samples were to be scored using a 0 (negative, no staining) to 3+ (brightest staining) scoring system for cytoplasmic and nuclear staining, and H- scores calculated using formula: 1x(percentage of cells stained 1+) + 2x(percentage of cells stained 2+) + 3x(percentage of cells stained 3+) .
Time Frame: Randomization, Cycle 2, end of study
Population: Zero participants were analyzed. The study was terminated and no data was collected.
Groups:
- Capecitabine + Enzastaurin: Capecitabine: 1250 milligrams per square meter (mg/m^2) twice daily (BID) on Days 1-14 followed by a 1-week rest period (Days 15-21) for each 21-day cycle until progressive disease.
  Enzastaurin: 1125-milligram (mg) loading dose on Day 1 of Cycle 1, then 500 mg daily on subsequent days to complete 21-day cycles until progressive disease.
- Capecitabine + Placebo: Capecitabine: 1250 mg/m^2 BID on Days 1-14 followed by a 1-week rest period (Days 15-21) for each 21-day cycle until progressive disease.
  Placebo: 4 tablets orally, daily, to complete 21-day cycles until progressive disease.
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve During One Dosing Interval at Steady State
Description: Area Under the Concentration versus time curve during 1 dosing interval at steady state (AUCτ,ss) for Cycle 2 Day 1 for Enzastaurin, its metabolite LY326020 and total analytes (enzastaurin + LY326020). AUCτ,ss was calculated using concentration versus time data by post hoc estimation of enzastaurin, its metabolite LY326020, and total analytes (enzastaurin + LY326020).
Time Frame: From pre-dose to 24 hours post-dose on Day 1 of Cycle 2
Population: All randomized participants who received at least 1 dose of enzastaurin and had data for AUCτ,ss analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles*hour per liter (nmol*hr/L)
Arm/Group | Capecitabine + Enzastaurin
Number analyzed (Participants) | 11
nanomoles*hour per liter (nmol*hr/L)
  Enzastaurin | 90000 (99)
  Enzastaurin Metabolite LY326020 | 40700 (31)
  Total Analytes (enzastaurin + LY326020) | 137000 (66)

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve Versus Time From Time 0 to Last Quantifiable Value (AUC0-tlast) of Capecitabine
Description: AUC0-tlast for Capecitabine, 5'-deoxy-5-fluorouridine (5'-DFUR) and 5-fluorouracil (5-FU) was calculated from the plasma concentration-time data for each analyte for Cycle 2, Day 1.
Time Frame: Pre-dose to 6 hours post-dose on Day 1 of Cycle 2
Population: All randomized participants who received at least 1 dose of capecitabine and had data for AUC 0-tlast analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliter (ug*hr/mL)
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo
Number analyzed (Participants) | 8 | 8
micrograms*hour/milliliter (ug*hr/mL)
  Capecitabine | 6.09 (57) | 4.18 (70)
  5'-deoxy-5-fluorouridine (5'-DFUR) | 11.6 (44) | 11.0 (31)
  5-fluorouracil (5-FU) | 0.683 (60) | 0.358 (42)

5. Secondary Outcome: Pharmacokinetics: Maximum Observed Concentration (Cmax) of Capecitabine
Description: Cmax for Capecitabine, 5'-deoxy-5-fluorouridine (5'-DFUR) and its metabolites 5-fluorouracil (5-FU) was calculated from the plasma concentration-time data for each analyte for Day 1 of Cycle 2.
Time Frame: From pre-dose to 6 hours post-dose on Day 1 of Cycle 2
Population: All randomized participants who received at least 1 dose of capecitabine and had data for Cmax analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter(ug/mL)
Groups:
- Capecitabine + Enzastaurin: Capecitabine: 1250 milligrams per square meter (mg/m^2), twice daily on Days 1-14 with a1 week rest period for 21-day cycles until progressive disease
  Enzastaurin: 1125 milligram (mg) loading dose on Day 1 of Cycle 1 and 500 mg daily on following days to complete 21-day cycles until progressive disease
- Capecitabine + Placebo: Capecitabine: 1250 mg/m^2, twice daily on Days 1-14 with a1 week rest period for 21-day cycles until progressive disease
  Placebo: taken as 4 oral tablets daily to complete 21-day cycles until progressive disease
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo
Number analyzed (Participants) | 8 | 8
micrograms/milliliter(ug/mL)
  Capecitabine | 4.42 (88) | 2.75 (114)
  5-DFUR | 6.09 (80) | 6.05 (69)
  5-FU | 0.374 (113) | 0.206 (73)

6. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Objective Response Rate)
Description: Response rate was defined as percent of participants with objective response [CR or PR] over randomized and treated participants using the Response Evaluation Criteria in Solid Tumors (RECIST v1.0) Guidelines. CR was defined as the disappearance of all tumor lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum of LDs or complete disappearance of target lesions, with persistence (but not worsening) of one or more non-target lesions. No new lesions may have appeared.
Time Frame: Randomization to last visit (up to 9.66 months)
Population: Intent-to-treat (ITT) population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Capecitabine + Enzastaurin: Capecitabine: 1250 milligrams per square meter (mg/m^2), twice daily on Days 1-14 with a1-week rest period for 21-day cycles until progressive disease
  Enzastaurin: 1125 milligram (mg) loading dose on Day 1 of Cycle 1 and 500 mg daily on following days to complete 21-day cycles until progressive disease
- Capecitabine + Placebo: Capecitabine: 1250 mg/m^2 twice daily on Days 1-14 with a1-week rest period for 21-day cycles until progressive disease
  Placebo: taken as 4 oral tablets daily to complete 21-day cycles until progressive disease
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo
Number analyzed (Participants) | 42 | 43
percentage of participants | 11.9 [4 to 26] | 11.6 [4 to 25]
Statistical Analysis 1: Comparison: Capecitabine + Enzastaurin vs Capecitabine + Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact — 1-sided significance level was 0.20

7. Secondary Outcome: Duration of Response (DOR)
Description: The DOR was defined as the time from first objective status assessment of complete response (CR) or partial response (PR) to the first time of progression or death as a result of any cause. According to the Response Evaluation Criteria in Solid Tumors (RECIST V1.0) criteria, CR was the disappearance of all tumor lesions. PR was at least a 30% decrease in the sum of the longest diameter (LD) of target lesions or complete disappearance of target lesions, with persistence (but not worsening) of 1 or more non-target lesions, with occurrence of no new lesions. For participants not known to have died as of the data cut-off date and who did not have progressive disease, DOR was censored at the date of last visit with adequate assessment. For participants who received subsequent anticancer therapy (after discontinuation from the study treatment) prior to disease progression or death, DOR was censored at the date of last visit with adequate assessment.
Time Frame: Randomization to last visit (up to 9.66 months)
Population: Intent to treat (ITT) population: All randomized participants who received at least 1 dose of study drug with a CR or PR. Participants censored: Capecitabine + Enzastaurin = 3; Capecitabine + Placebo = 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo
Number analyzed (Participants) | 5 | 5
months | 4.27 [2.17 to 4.27] | 3.47 [2.79 to NA] — Not evaluable due to too few data points.
Statistical Analysis 1: Comparison: Capecitabine + Enzastaurin vs Capecitabine + Placebo; Test type: Superiority or Other; p = 0.812, Log Rank

8. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time in months from the date of study enrollment to the date of death from any cause. For participants not known to have died as of the cut-off date, OS was censored at the last contact date.
Time Frame: Randomization to date of death from any cause up to 20.83 months
Population: Intent-to-treat (ITT) population: All randomized participants who received at least 1 dose of study drug. Participants censored: Capecitabine + Enzastaurin = 23; Capecitabine + Placebo = 28.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo
Number analyzed (Participants) | 42 | 43
months | 9.86 [7.03 to 16.59] | 14.88 [9.86 to 19.32]
Statistical Analysis 1: Comparison: Capecitabine + Enzastaurin vs Capecitabine + Placebo; Test type: Superiority or Other; p = 0.181, Log Rank

9. Secondary Outcome: Pharmacology Toxicity and Adverse Events (AEs)
Description: Data presented are the number of participants who experienced serious AEs, AEs, death due to progressive disease (PD), death due to AEs while on treatment and death during the 30-day post-treatment. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion [Cycle 19 (21 days/cycle) and 30-day safety follow-up]
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine + Enzastaurin | Capecitabine + Placebo
Number analyzed (Participants) | 42 | 43
Participants
  Serious AEs | 12 | 12
  Other non-serious AEs | 38 | 40
  Deaths Due to PD | 13 | 12
  Deaths Due to AEs | 4 | 2
  Deaths in 30-day follow-up | 6 | 1

ADVERSE EVENTS:
Time Frame: Baseline to study completion [Cycle 19 (21 days/cycle) and 30-day safety follow-up]
Description: Study-specific clinical outcomes due to progressive disease (PD) were not considered to be serious adverse events (SAEs) unless it was deemed related to study drug by the investigator.
Groups:
- A - Capecitabine + Enzastaurin: Capecitabine: 1250 milligrams per square meter (mg/m^2) twice daily (BID) on Days 1-14 followed by a 1-week rest period (Days 15-21) for each 21-day cycle until progressive disease.
  Enzastaurin: 1125-milligram (mg) loading dose on Day 1 of Cycle 1, then 500 mg daily on subsequent days to complete 21-day cycles until progressive disease.
- B - Capecitabine + Placebo: Capecitabine: 1250 mg/m^2 BID on Days 1-14 followed by a 1-week rest period (Days 15-21) for each 21-day cycle until progressive disease.
  Placebo: 4 tablets orally, daily, to complete 21-day cycles until progressive disease.
Arm/Group | A - Capecitabine + Enzastaurin | B - Capecitabine + Placebo
Serious Adverse Events (participants affected / at risk) | 12/42 | 12/43
Other Adverse Events (participants affected / at risk) | 38/42 | 40/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Capecitabine + Enzastaurin (N=42) | B - Capecitabine + Placebo (N=43)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Biopsy (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - Capecitabine + Enzastaurin (N=42) | B - Capecitabine + Placebo (N=43)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (5) | 1 (2)
Lacrimation increased (Eye disorders) | 1 (1) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 20 (27) | 17 (24)
Nausea (Gastrointestinal disorders) | 17 (23) | 21 (27)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 3 (4)
Vomiting (Gastrointestinal disorders) | 13 (18) | 18 (24)
Asthenia (General disorders) | 3 (3) | 2 (3)
Fatigue (General disorders) | 13 (13) | 14 (14)
Influenza like illness (General disorders) | 2 (2) | 3 (3)
Mucosal inflammation (General disorders) | 5 (6) | 2 (3)
Oedema peripheral (General disorders) | 7 (7) | 3 (5)
Pain (General disorders) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (5)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3) | 0 (0)
Haemoglobin decreased (Investigations) | 4 (5) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (5) | 1 (1)
Urine colour abnormal (Investigations) | 6 (6) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 12 (13) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (9)
Dizziness (Nervous system disorders) | 7 (7) | 7 (13)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (25) | 18 (20)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (9)
Skin reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days